CLINICAL TRIAL: NCT05005897
Title: Vitamin B12 Status in Infancy and the Effect of Providing Vitamin B12 to Infants With Signs of Suboptimal Vitamin B12 Status - a Registry-based, Randomized Controlled Trial
Brief Title: Early Infant Micronutrition and Development
Acronym: RART
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: University of Bergen (Other); University of Oslo (Other); Inland Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9305-150426; U1111-1267-0112 (Other: World Health Organization)
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Vitamin B 12 Deficiency
Keywords: Nutrition; Vitamins; Breastfeeding; Infant; Neurodevelopment; Growth; Clinical trial
MeSH Terms: conditions — Vitamin B 12 Deficiency; Breast Feeding | interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening - treatment (Experimental): From 6 weeks of age, infants will be screened for elevated plasma total homocysteine concentrations. Those who have a concentration above the defined cut-off will be treated with cobalamin (vitamin B12).
  Interventions: Biological: Cyanocobalamin
- Control (No Intervention): The control-group sample will be stored and analyzed when the child is 12 months old. Those with elevated tHcy will contribute to the control group.

INTERVENTIONS:
Biological: Cyanocobalamin — Intramuscular injection of 400 µg cobalamin to children with elevated thcy at enrollment
  Other Names: Vitamin B12
  Arms: Screening - treatment

SUMMARY:
Globally, vitamin B12 deficiency is one of the most common micronutrient deficiencies. Poor status is also seen in affluent countries such as in Norway. Vitamin B12 is crucial for normal cell division and differentiation and necessary for the development and myelination of the central nervous system. Deficiency is also associated with impaired fetal and infant growth. In the proposed study we will measure the effect of daily oral vitamin B12 supplementation infants on neurodevelopment. We also aim to measure the impact of B12 supplementation on several other outcomes.

Study design: Individually randomized double-blind placebo-controlled trial breastfed infants who will be assigned to a screening group (in which measurements will be obtained immediately) or a control group (in which serum will be stored and measurements done after one year).

Pregnant women will be informed about the study during their first antenatal visit at the clinic and that we will re-approach them on their 6-week visit to their public health nurse. Infants who are deficient will be treated with peroral or intramuscular injections with 400 µg cyano-cobalamin.

Infants in the control group will not be offered any intervention their blood sample will be stored for one year and then analyzed for the same nutrients as the intervention group.

Outcomes: Primary: (i) neurodevelopment in children measured at 12 months of age (ii) growth in children measured by attained weight and length at 12 months. Secondary: (i) neurodevelopment and cognitive functioning in children later in life

ELIGIBILITY:
Inclusion Criteria:

1. Availability of informed verbal consent
2. Plan to reside in the defined study area for the next 12 months
3. Mothers intend to breastfeed their children for at least 8 months, and exclusively for 4 months

Exclusion Criteria:

1. Severe systemic illness requiring hospitalization
2. Growth retardation
3. Severe congenital malformations
4. Plasma cobalamin concentration <148 pmol/L (These children will be treated for vitamin B12 deficiency and not included in the RCT, but will be included in the cohort design)

Ages: 1 Month to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopment | 12 months of age
  Bayley Scales of Infant Development 4th edition
Prevalence of vitamin B12 deficiency | 1-3 months of age
  Number of children with elevated plasma homocysteine or low cobalamin
Prevalence of other vitamin deficiencies | 1-3 months of age
  Number of infants with vitamin deficiencies other than vitamin B12 deficiency

SECONDARY OUTCOMES:
Neurodevelopment measured by the Ages and Stages Questionaire | 4-12 months of age
  Ages and Stages Questionnaire version 3 repeated throughout infancy
Vagal tone | 12 months of age
  Heart rate variability
Eye tracking | 12 months of age
  Visual acuity, visuospatial orientation, and attention to social cues
Neurodevelopment later in childhood | 5 years
  General cognitive abilities ("IQ") assessed by the Wechsler Preschool and Primary Scale of Intelligence
Adverse events | 3 months after treatment with vitamin B12
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
Thyroid function | 12 months of age
  Infant thyroid function measured by the concentration of the hormones TSH, T3, and T4

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Strand, M.D. / Ph.D., Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available not later than 5 years after the study have completed enrollment and the first year of follow-up of all children.
Access Criteria: Data available on request. In order to meet ethical requirements for the use of confidential patient data, requests must be approved by Regional Committee for Medical and Health Research Ethics in Norway.

REFERENCES:
- [Background] Hay G, Johnston C, Whitelaw A, Trygg K, Refsum H. Folate and cobalamin status in relation to breastfeeding and weaning in healthy infants. Am J Clin Nutr. 2008 Jul;88(1):105-14. doi: 10.1093/ajcn/88.1.105. PMID 18614730
- [Background] Torsvik I, Ueland PM, Markestad T, Bjorke-Monsen AL. Cobalamin supplementation improves motor development and regurgitations in infants: results from a randomized intervention study. Am J Clin Nutr. 2013 Nov;98(5):1233-40. doi: 10.3945/ajcn.113.061549. Epub 2013 Sep 11. PMID 24025626
- [Background] Dror DK, Allen LH. Effect of vitamin B12 deficiency on neurodevelopment in infants: current knowledge and possible mechanisms. Nutr Rev. 2008 May;66(5):250-5. doi: 10.1111/j.1753-4887.2008.00031.x. PMID 18454811
- [Background] Kvestad I, Taneja S, Kumar T, Hysing M, Refsum H, Yajnik CS, Bhandari N, Strand TA; Folate and Vitamin B12 Study Group. Vitamin B12 and Folic Acid Improve Gross Motor and Problem-Solving Skills in Young North Indian Children: A Randomized Placebo-Controlled Trial. PLoS One. 2015 Jun 22;10(6):e0129915. doi: 10.1371/journal.pone.0129915. eCollection 2015. PMID 26098427
- [Background] Bjorke-Monsen AL. Is exclusive breastfeeding ensuring an optimal micronutrient status and psychomotor development in infants? Clin Biochem. 2014 Jun;47(9):714. doi: 10.1016/j.clinbiochem.2014.05.022. Epub 2014 May 17. No abstract available. PMID 24845709
- [Background] Forssman L, Ashorn P, Ashorn U, Maleta K, Matchado A, Kortekangas E, Leppanen JM. Eye-tracking-based assessment of cognitive function in low-resource settings. Arch Dis Child. 2017 Apr;102(4):301-302. doi: 10.1136/archdischild-2016-310525. Epub 2016 Aug 22. PMID 27551061
- [Background] Graziano P, Derefinko K. Cardiac vagal control and children's adaptive functioning: a meta-analysis. Biol Psychol. 2013 Sep;94(1):22-37. doi: 10.1016/j.biopsycho.2013.04.011. Epub 2013 May 4. PMID 23648264
- [Background] Strand TA, Taneja S, Ueland PM, Refsum H, Bahl R, Schneede J, Sommerfelt H, Bhandari N. Cobalamin and folate status predicts mental development scores in North Indian children 12-18 mo of age. Am J Clin Nutr. 2013 Feb;97(2):310-7. doi: 10.3945/ajcn.111.032268. Epub 2013 Jan 2. PMID 23283502
- [Derived] Bjorkevoll SMG, O'Keeffe M, Konijnenberg C, Solvik BS, Sodal AF, Kaldenbach S, McCann A, Ueland PM, Kvestad I, Ersvaer E, Holten-Andersen MN, Bakken KS, Strand TA. Infant vitamin B12 status and its predictors - cross-sectional baseline results from an ongoing randomized controlled trial. Am J Clin Nutr. 2025 Sep;122(3):803-810. doi: 10.1016/j.ajcnut.2025.06.029. Epub 2025 Jul 1. PMID 40609749
- [Derived] Bakken KS, Kvestad I, Bjorkevoll SMG, Solvik BS, Kaldenbach S, McCann A, Holten-Andersen MN, Ersvaer E, Konijnenberg C, Strand TA. Vitamin B12 status in infancy and the effect of a vitamin B12 injection in infants with subclinical vitamin B12 deficiency: study protocol for a register-based randomised controlled trial. BMJ Open. 2023 Apr 20;13(4):e069102. doi: 10.1136/bmjopen-2022-069102. PMID 37080624